CLINICAL TRIAL: NCT00002452
Title: A Multicenter, Open-Label, Pilot Study to Evaluate the Safety and Activity of L-756423/Indinavir Sulfate, 800/400 Mg b.i.d. in Combination With Two nRTIs in HIV-Infected Patients Who Failed an Indinavir Containing Regimen
Brief Title: A Study on the Safety and Effectiveness of L-756423 Plus Indinavir in HIV-Positive Patients Who Have Previously Taken Indinavir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 300A; 008-00
Record Dates: First submitted 2000-01-17; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Indinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — L 756423; Indinavir

INTERVENTIONS:
Drug: L-756423
Drug: Indinavir sulfate

SUMMARY:
The purpose of this study is to see if L-756423, an anti-HIV drug, is safe to give with indinavir and if it works well at lowering the level of HIV in the blood (viral load).

DETAILED DESCRIPTION:
All patients receive L-756423 plus indinavir plus two licensed nucleoside reverse transcriptase inhibitors (NRTIs), at least one to which the patient is naive. Patients remain on the drug regimen for 12 weeks (with possible extension to 16 weeks). Patients are evaluated with physical examinations and laboratory tests for blood and urine at Weeks 1, 2, 4, 6, 8, and 12 and two weeks post study. Plasma viral RNA is measured at Weeks 1, 2, 4, 6, 8, and 12. CD4 cell counts are measured at Weeks 2,4,8, and 12.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Are at least 18 years old.
* Have a viral load of at least 1,000 copies/ml.
* Have a CD4 cell count of at least 100 cells/mm3.
* Have experienced treatment failure (your viral load increased significantly) within 24 weeks of study entry while taking indinavir.

Exclusion Criteria

You will not be eligible for this study if you:

* Are taking nonnucleoside reverse transcriptase inhibitors (NNRTIs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Georgetown Univ, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Hawaii AIDS Clinical Trial Unit, Honolulu, Hawaii
  - The CORE Ctr, Chicago, Illinois
  - Cornell Clinical Trials Unit - Chelsea Clinic, New York, New York
  - Pittsburgh Treatment Ctr / Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee